CLINICAL TRIAL: NCT00221377
Title: "Cuffed Versus Uncuffed Tracheal Tubes in Small Children"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STV1/05; no grants
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2011-12

CONDITIONS: Need for Tracheal Tube Exchange; Presence of Post-extubation Laryngeal Oedema
Keywords: intubation; trachea; tube; cuff; children
MeSH Terms: conditions — Tracheal Diseases

INTERVENTIONS:
Device: Intubation using tracheal tubes with or without cuff

SUMMARY:
This randomized controlled multi-centre trial in children from birth up to < 5 years of age aims to demonstrate equivalence as to the major outcome of post-extubation airway injury (stridor) comparing uncuffed tracheal tubes to current tracheal tubes with modern high volume - low pressure cuff combined with a cuff pressure release valve.

DETAILED DESCRIPTION:
The use of cuffed tracheal tubes is a controversial topic in paediatric anaesthesia and intensive care medicine. Cuffed tubes have traditionally been recommended for children older than 8 to 10 years. During the past decade, however, several authors have argued for the use of cuffed tracheal tubes in younger children and infants. A frequently cited argument against their use is the fear from post-extubation morbidity, allegedly caused by cuff induced tracheal and laryngeal airway injury. Using modern improved designed cuffed tracheal tubes, data from randomised prospective studies, performed in paediatric anaesthesia and intensive care units, suggest that using cuffed tracheal tubes do not carry an increased risk for airway morbidity as compared to uncuffed tracheal tubes in children below 8 years of age if correctly used. However, all these studies are based on single-centre experiences and/or included only a few neonates, infants and small children. Hence, there is equipoise as to the question, whether cuffed tubes are preferable over uncuffed standard tubes.

So, this randomized controlled multi-centre trial in children from birth up to < 5 years of age aims to demonstrate equivalence as to the major outcome of post-extubation airway injury (stridor) comparing uncuffed tracheal tubes to current tracheal tubes with modern high volume - low pressure cuff combined with a cuff pressure release valve.

The primary hypothesis relates to the main outcome criteria of this study, which is post-extubation morbidity as measured by the presence or absence of stridor after tracheal extubation. The null-hypothesis Ho is defined as no difference in the incidence rates of post-extubation morbidity between cuffed and uncuffed groups. The null-hypothesis (Ho: u-Diff = 0) will be compared with the alternative hypothesis (H1: u-Diff <> 0). The study is designed to detect a clinically unacceptable deterioration of 1.5% above the baseline airway-injury rate of 2.5% when using uncuffed tubes with a power of 90% and a type I error probability of less than 5%.

ELIGIBILITY:
Inclusion Criteria:

* Children aged from birth (weighing > 3 kg) to <5 years
* Children requiring oro-tracheal or naso-tracheal intubation with a Magil shaped tracheal tube or preformed (RAE) tracheal tube as a part of their anaesthetic care and planed IPPV during the surgical / interventional / diagnostic procedure
* Tracheal intubation performed using direct laryngoscopy
* Extubation after the procedure in the OR theatre
* Procedure performed in supine position
* Patients for elective and emergency surgery and/or interventions if there is no risk for regurgitation or pulmonary aspiration
* ASA I and II patients
* Written parental consent

Exclusion Criteria:

* No parental written consent obtained
* Known airway anomalies (airway stenosis, including Down's Syndrome)
* Known or suspected difficult intubation
* Known need for abnormal tube size
* Full stomach and/or at risk for regurgitation
* Surgery of the larynx and/or of the trachea and/or neck and/or upper oesophagus
* Pulmonary diseases (concurrent pneumonia or bronchial infection, asthma requiring inhalation medication, pulmonary malformations)
* ASA class III and higher
* Fiberoptic intubation or alternative intubation technique
* Patients planned for postoperative ventilation in the ICU
* Weight and/or height percentiles < 3% / > 97%

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4000 (Estimated)
Dates: Start 2005-04; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
post-extubation stridor (airway stenosis)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Weiss, Prof MD, Principal Investigator — University Children's Hospital, Anesthesiology
Locations (24):
- Anesthesia And Critical Care Medicine - Medical University, Innsbruck, Austria
- Departement of Anaesthesia - Cliniques Universitaire St. Luc, Brussels, Belgium
- Dept. of Anaesthesia and Reanimation - University Hospital Motol, Prague, Czechia
- Germany (8):
  - Klinik für Anasthesiologie und Operative Intensivmedizin - Klinikum Augsburg, Augsburg
  - Clinic of Anesthesiology - Charite-Universitätsmedizin, Berlin
  - Dep. Anesthesiology and Intensive Care - Helios Klinikum Berlin-Buch, Berlin
  - Dept. of Anaesthesia - Kinderkrankenhaus auf der Bult, Hanover
  - Dept. of Anaesthesia Kliniken Loerrach, Loerrach
  - Anaesthesia and Intensive Care - University Hospital Mannheim, Mannheim
  - Klinik für Anaesthesie, LMU München - Dr. U. Haunersches Kinderspital, München
  - Anaesthesia - Klinik St. Hedwig, Regensburg
- Slovakia (2):
  - Children's University Hospital - Dept. of Anaesthesia and Intensive Care, Bratislava
  - Dept. of Anaesthesia and Intensive Care - Faculty Hospital of Luis Pasteur, Košice
- Dept. of Anaesthesia and Intensive Care - Astrid Lindgrens Children's Hospital, Stockholm, Sweden
- Switzerland (6):
  - University Children's Hospital, Zurich, Canton of Zurich
  - Klinik für Anästhesie und Op. Intensivmedizin, Aarau
  - Klinik für Anästhesiologie - Inselspital, Bern
  - Dept. of Anaesthesia, Geneva Children's Hospital, Geneva
  - Service d'Anesthesiologie - CHUV, Lausanne
  - Anästhesie - Ostschweizer Kinderspital, Sankt Gallen
- United Kingdom (4):
  - Anaesthetics - Royal Aberdeen Children's Hospital, Aberdeen
  - Anaesthetic Department - Royal Hospital for Sick Children, Glasgow
  - Anaesthetic Department - Ledds General Infirmary, Leeds
  - Anaesthesia - Chelsa and Westminster NHS Trust, London